CLINICAL TRIAL: NCT05305781
Title: Prevalence and Epidemiology of Extra Renal Replacement Therapy
Brief Title: Study of the Determinants of Emergency Dialysis in Reunion Island
Acronym: PEPER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/CHU/24
Record Dates: First submitted 2022-02-28; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Dialysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Among patients followed by nephrologists, the frequency of emergency dialysis starts' and their social and clinical determinants are not well known, especially in Reunion Island. In this context, we aim to study and understand the determinants of emergency dialysis initiation. For Reunion Island, the data remain very fragmented.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥18 years
* Starting dialysis in a dialysis centre in Réunion Island
* Having expressed their non-opposition or Emergency inclusion (non-opposition collected afterwards)

Exclusion Criteria:

* Under legal protection (safeguard of justice, guardianship)
* Unable to answer questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We plan to include 200 newly dialysis patients in a year from the dialysis centres covering the major part of the Reunion Island.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Characteristics of emergency analysis | 24 hours
  Incidence rate of emergency dialysis

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Réunion, Saint-Denis, Reunion